CLINICAL TRIAL: NCT05167435
Title: Myofascial Release Technique vs Posterior-anterior Glide on Non-specific Low Back Pain: a Randomized Controlled Trial
Brief Title: Myofascial Release Technique vs Posterior-anterior Glide on Non-specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Syeda Waniya Riaz, Syeda Waniya Riaz, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Swaniya
Record Dates: First submitted 2021-11-25; First posted 2021-12-22 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Low Back Pain
Keywords: Chronic Pain; Disabled Persons; Myofascial Release; Low back pain; Back pain; Exercise Therapy; Quality of life
MeSH Terms: conditions — Low Back Pain; Chronic Pain; Back Pain

STUDY DESIGN:
Intervention Model Description: It is a randomized controlled trial. Total 80 patients will be recruited, 40 in each group that includes 4 patients as a dropout in both groups. There will be one interventional group and one control group. Treatment will be allocated using a random number sheet generated by SPSS software version 21. Participants are assigned to one of two groups in parallel for the duration of the study.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor involved in the clinical trial will be prevented from having knowledge of the interventions assigned to individual participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Intervention) (Experimental): Myofascial release (Following Cross-hand release techniques of myofascial release in a manner of 2 minutes approach:
  Cross-Hand Release of Back [For Thoracolumbar Fascia] Cross-Hand Release of the Lumbosacral Junction [L5-S1] Cross-Hand Release of Lateral low back area [for quadratus lumborum]) will be provided with conventional therapy including stretching exercises (Stretching of Latissimus Dorsi [10 seconds hold, 10 reps, 2 sets], Quadratus Lumborum Stretching [10 seconds hold, 3 reps, 1 set bilaterally], Lower Back Stretching [10 seconds hold, 10 reps, 2 sets], Hamstring Stretching [10 seconds hold, 10 reps, 2 sets bilaterally], Tensor Fasciae Latae Stretching [10 sec hold, 10 reps, 2 sets bilaterally] with duration rest will be of thirty seconds after five minutes) and Thermotherapy will be given for 20 minutes
  Interventions: Other: Myofascial Release Experimental
- Group B (Control) (Active Comparator): Posterior-anterior glide: Grade 1-4 [depending on tolerance] (120 oscillations per minute x 3 sets, Duration of rest between each set: 30 seconds) will be provided with the same conventional therapy as in Group A (Intervention)
  Interventions: Other: Posterior-Anterior Glide

INTERVENTIONS:
Other: Myofascial Release Experimental — Myofascial release is a gentle sustained pressure that elongates fascial adhesions so that tissue can return to proper realignment.
  Arms: Group A (Intervention)
Other: Posterior-Anterior Glide — Posterior-anterior mobilization is a standard assessment and treatment technique for most clinicians. It is a mobilization technique that involves passive oscillatory movements applied to a vertebral segment in a posteroanterior direction (Back to front).
  Arms: Group B (Control)

SUMMARY:
The objective of this randomized control trial is to determine the effectiveness of myofascial release in patients with nonspecific low back pain to improve Pain, Disability, and Quality of life This study is being conducted at the Outpatient Physiotherapy department of Sindh Institute of Physical Medicine and Rehabilitation, Karachi (former institute of Dow University of Health Sciences) and Musculoskeletal outpatient department of Dr. Ruth K. M. Pfau, Civil Hospital Karachi among 72 patients with nonspecific back pain on the basis of non-probability purposive sample technique with screening for study criteria through a consultant physician (blinded). After taking informed consent, all participants will be randomly allocated into two groups through a second researcher who is not involved in screening, baseline assessment, and providing intervention. Group 1 will receive myofascial release with generalized low back stretching and thermotherapy and Group 2 will receive Posterior-anterior glide with generalized low back stretching and thermotherapy. A total of 18 sessions will be provided. Outcomes will be assessed at baseline, at the last session, and after 12 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

Nonspecific low back pain > 3 months

8 and 45 years of age

IPMR and civil musculoskeletal outpatient department patients

Without referred leg pain

Exclusion Criteria:

Any trauma, spinal infection or tumor, spinal fracture, previous spinal surgery, systemic disease, fibromyalgia, cauda equine syndrome, serious chronic disease, specific neurological disease (stroke, MS, and Parkinson's disease)

Uncontrolled diabetes or hypertension

Pregnant females

Spondylolisthesis, spinal stenosis, spondylolysis, ankylosing spondylitis, structural deformity, congenital deformation, disc disease, sacroiliitis, severe structural deformity, scoliosis, active structural deficit, and severe postural abnormality

Acute coronary disease

Asthmatic patients

Any contraindication prescribed for myofascial treatment

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain on Short Form McGill Questionnaire 2 (SFMPQ-2) at 6 weeks (post intervention). | Baseline and Post Intervention
  The patient will be asked to mark the Quality and Intensity of pain on a scale of 0-10 that measures the level of pain. The 0 refers no pain and 10 refers worse possible pain and perceived as maximum.
Change from baseline in pain on Short Form McGill Questionnaire 2 (SFMPQ-2) at 12 weeks follow-up. | Baseline and 12 weeks follow-up
  The patient will be asked to mark the Quality and Intensity of pain on a scale of 0-10 that measures the level of pain. The 0 refers no pain and 10 refers worse possible pain and perceived as maximum.
Change from 6 weeks (post intervention) in pain on Short Form McGill Questionnaire 2 (SFMPQ-2) at 12 weeks follow-up. | Post Intervention and 12 weeks follow-up
  The patient will be asked to mark the Quality and Intensity of pain on a scale of 0-10 that measures the level of pain. The 0 refers no pain and 10 refers worse possible pain and perceived as maximum.
Change from baseline in disability on the Roland Morris Disability Questionnaire at 6 weeks (post intervention).. | Baseline and Post Intervention
  A list of 24 sentences will be provided that are found to be difficult to be done by back pain patients. The patient will be asked to mark the sentence. The higher the number of sentences represents the greater intensity of disability means extreme disability. On the other hand the lower the number of sentences marked means the lower the score on the scale for example like 0 (zero) shows no disability.
Change from baseline in disability on the Roland Morris Disability Questionnaire at 12 weeks follow-up. | Baseline and 12 weeks follow-up
  A list of 24 sentences will be provided that are found to be difficult to be done by back pain patients. The patient will be asked to mark the sentence. The higher the number of sentences represents the greater intensity of disability means extreme disability. On the other hand the lower the number of sentences marked means the lower the score on the scale for example like 0 (zero) shows no disability.
Change from 6 weeks (post intervention) in disability on the Roland Morris Disability Questionnaire at 12 weeks follow-up. | Post Intervention and 12 weeks follow-up
  A list of 24 sentences will be provided that are found to be difficult to be done by back pain patients. The patient will be asked to mark the sentence. The higher the number of sentences represents the greater intensity of disability means extreme disability. On the other hand the lower the number of sentences marked means the lower the score on the scale for example like 0 (zero) shows no disability.
Change from baseline in Quality of life on the WHOQOL BREF at 6 weeks (post intervention). | Baseline and Post Intervention
  This questionnaire assess the quality of life within the context of an individual's physical health, psychological, social relationships and environment. Other than these 4 domains 2 questions are asked separately to evaluate an individuals overall perception of quality of life and about an individuals overall perception of their health. The higher the score denote the higher the quality of life and lower score denotes lower quality of life. All 26 assessment questions in the questionnaire has a range of 1-5. 3 of the questions are negatively phrased and so are reversed scored when calculating the domain scores - a score of 5 becomes a 1 and vice versa, a score of 4 becomes a two and vice versa etc. This is performed on questions 3, 4, and 26. You do this before calculating any domain scores. The domain scores are than added to get the final score.
Change from baseline in Quality of life on the WHOQOL BREF at 12 weeks follow-up. | Baseline and 12 weeks follow-up
  This questionnaire assess the quality of life within the context of an individual's physical health, psychological, social relationships and environment. Other than these 4 domains 2 questions are asked separately to evaluate an individuals overall perception of quality of life and about an individuals overall perception of their health. The higher the score denote the higher the quality of life and lower score denotes lower quality of life. All 26 assessment questions in the questionnaire has a range of 1-5. 3 of the questions are negatively phrased and so are reversed scored when calculating the domain scores - a score of 5 becomes a 1 and vice versa, a score of 4 becomes a two and vice versa etc. This is performed on questions 3, 4, and 26. You do this before calculating any domain scores. The domain scores are than added to get the final score.
Change from 6 weeks (post intervention) in Quality of life on the WHOQOL BREF at 12 weeks follow-up. | Post Intervention and 12 weeks follow-up
  This questionnaire assess the quality of life within the context of an individual's physical health, psychological, social relationships and environment. Other than these 4 domains 2 questions are asked separately to evaluate an individuals overall perception of quality of life and about an individuals overall perception of their health. The higher the score denote the higher the quality of life and lower score denotes lower quality of life. All 26 assessment questions in the questionnaire has a range of 1-5. 3 of the questions are negatively phrased and so are reversed scored when calculating the domain scores - a score of 5 becomes a 1 and vice versa, a score of 4 becomes a two and vice versa etc. This is performed on questions 3, 4, and 26. You do this before calculating any domain scores. The domain scores are than added to get the final score.

CONTACTS AND LOCATIONS:
Locations (3):
- Pakistan (3):
  - Dow University of Health Sciences, Karachi, Sindh
  - Dr. Ruth.K.M.Pfau Civil Hospital, Karachi, Sindh
  - Sindh Institute o Physical Medicine and Rehabilitation, Karachi, Sindh

REFERENCES:
- [Background] Blyth FM, Noguchi N. Chronic musculoskeletal pain and its impact on older people. Best Pract Res Clin Rheumatol. 2017 Apr;31(2):160-168. doi: 10.1016/j.berh.2017.10.004. Epub 2017 Nov 4. PMID 29224694
- [Background] Chenot JF, Greitemann B, Kladny B, Petzke F, Pfingsten M, Schorr SG. Non-Specific Low Back Pain. Dtsch Arztebl Int. 2017 Dec 25;114(51-52):883-890. doi: 10.3238/arztebl.2017.0883. PMID 29321099
- [Background] Ehrlich GE. Low back pain. Bull World Health Organ. 2003;81(9):671-6. Epub 2003 Nov 14. PMID 14710509
- [Background] Savigny P, Watson P, Underwood M; Guideline Development Group. Early management of persistent non-specific low back pain: summary of NICE guidance. BMJ. 2009 Jun 4;338:b1805. doi: 10.1136/bmj.b1805. No abstract available. PMID 19502217
- [Background] Walker J. Back pain: pathogenesis, diagnosis and management. Nurs Stand. 2012 Dec 5-11;27(14):49-56; quiz 58. doi: 10.7748/ns2012.12.27.14.49.c9478. PMID 23488026
- [Background] Hoy D, Brooks P, Blyth F, Buchbinder R. The Epidemiology of low back pain. Best Pract Res Clin Rheumatol. 2010 Dec;24(6):769-81. doi: 10.1016/j.berh.2010.10.002. PMID 21665125
- [Background] Arguisuelas MD, Lison JF, Sanchez-Zuriaga D, Martinez-Hurtado I, Domenech-Fernandez J. Effects of Myofascial Release in Nonspecific Chronic Low Back Pain: A Randomized Clinical Trial. Spine (Phila Pa 1976). 2017 May 1;42(9):627-634. doi: 10.1097/BRS.0000000000001897. PMID 28441294
- [Background] Laimi K, Makila A, Barlund E, Katajapuu N, Oksanen A, Seikkula V, Karppinen J, Saltychev M. Effectiveness of myofascial release in treatment of chronic musculoskeletal pain: a systematic review. Clin Rehabil. 2018 Apr;32(4):440-450. doi: 10.1177/0269215517732820. Epub 2017 Sep 28. PMID 28956477
- [Background] Husky MM, Ferdous Farin F, Compagnone P, Fermanian C, Kovess-Masfety V. Chronic back pain and its association with quality of life in a large French population survey. Health Qual Life Outcomes. 2018 Sep 26;16(1):195. doi: 10.1186/s12955-018-1018-4. PMID 30257670
- [Background] Ajimsha MS, Al-Mudahka NR, Al-Madzhar JA. Effectiveness of myofascial release: systematic review of randomized controlled trials. J Bodyw Mov Ther. 2015 Jan;19(1):102-12. doi: 10.1016/j.jbmt.2014.06.001. Epub 2014 Jun 13. PMID 25603749
- [Background] Yu SH, Sim YH, Kim MH, Bang JH, Son KH, Kim JW, Kim HJ. The effect of abdominal drawing-in exercise and myofascial release on pain, flexibility, and balance of elderly females. J Phys Ther Sci. 2016 Oct;28(10):2812-2815. doi: 10.1589/jpts.28.2812. Epub 2016 Oct 28. PMID 27821941
- [Background] Buchbinder R, Blyth FM, March LM, Brooks P, Woolf AD, Hoy DG. Placing the global burden of low back pain in context. Best Pract Res Clin Rheumatol. 2013 Oct;27(5):575-89. doi: 10.1016/j.berh.2013.10.007. Epub 2013 Oct 12. PMID 24315140
- [Background] Fouquet N, Bodin J, Descatha A, Petit A, Ramond A, Ha C, Roquelaure Y. Prevalence of thoracic spine pain in a surveillance network. Occup Med (Lond). 2015 Mar;65(2):122-5. doi: 10.1093/occmed/kqu151. Epub 2014 Oct 24. PMID 25344959
- [Background] Roland M, Fairbank J. The Roland-Morris Disability Questionnaire and the Oswestry Disability Questionnaire. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3115-24. doi: 10.1097/00007632-200012150-00006. No abstract available. PMID 11124727
- [Background] Dworkin RH, Turk DC, Trudeau JJ, Benson C, Biondi DM, Katz NP, Kim M. Validation of the Short-form McGill Pain Questionnaire-2 (SF-MPQ-2) in acute low back pain. J Pain. 2015 Apr;16(4):357-66. doi: 10.1016/j.jpain.2015.01.012. Epub 2015 Jan 29. PMID 25640290
- [Background] Nadler SF, Weingand K, Kruse RJ. The physiologic basis and clinical applications of cryotherapy and thermotherapy for the pain practitioner. Pain Physician. 2004 Jul;7(3):395-9. PMID 16858479
- [Background] Qaseem A, Wilt TJ, McLean RM, Forciea MA; Clinical Guidelines Committee of the American College of Physicians; Denberg TD, Barry MJ, Boyd C, Chow RD, Fitterman N, Harris RP, Humphrey LL, Vijan S. Noninvasive Treatments for Acute, Subacute, and Chronic Low Back Pain: A Clinical Practice Guideline From the American College of Physicians. Ann Intern Med. 2017 Apr 4;166(7):514-530. doi: 10.7326/M16-2367. Epub 2017 Feb 14. PMID 28192789
- [Background] Baig AAM, Ahmed SI, Ali SS, Rahmani A, Siddiqui F. Role of posterior-anterior vertebral mobilization versus thermotherapy in non specific lower back pain. Pak J Med Sci. 2018 Mar-Apr;34(2):435-439. doi: 10.12669/pjms.342.12402. PMID 29805422
- [Background] Bernstein IA, Malik Q, Carville S, Ward S. Low back pain and sciatica: summary of NICE guidance. BMJ. 2017 Jan 6;356:i6748. doi: 10.1136/bmj.i6748. No abstract available. PMID 28062522
- [Background] Anderson RU, Wise D, Sawyer T, Glowe P, Orenberg EK. 6-day intensive treatment protocol for refractory chronic prostatitis/chronic pelvic pain syndrome using myofascial release and paradoxical relaxation training. J Urol. 2011 Apr;185(4):1294-9. doi: 10.1016/j.juro.2010.11.076. Epub 2011 Feb 22. PMID 21334027
- [Background] Hodges PW, Danneels L. Changes in Structure and Function of the Back Muscles in Low Back Pain: Different Time Points, Observations, and Mechanisms. J Orthop Sports Phys Ther. 2019 Jun;49(6):464-476. doi: 10.2519/jospt.2019.8827. PMID 31151377
- [Background] Goubert D, Oosterwijck JV, Meeus M, Danneels L. Structural Changes of Lumbar Muscles in Non-specific Low Back Pain: A Systematic Review. Pain Physician. 2016 Sep-Oct;19(7):E985-E1000. PMID 27676689
- [Background] Bae HI, Kim DY, Sung YH. Effects of a static stretch using a load on low back pain patients with shortened tensor fascia lata. J Exerc Rehabil. 2017 Apr 30;13(2):227-231. doi: 10.12965/jer.1734910.455. eCollection 2017 Apr. PMID 28503538
- See also: Doherty M, Ralston S.H. Musculoskeletal disease. Davidson's Principles and Practice of Medicine, 21st Edition. Churchill Livingstone, Elsevier. 2010. — https://www.elsevier.com/books/davidsons-principles-and-practice-of-medicine/ralston/978-0-7020-7028-0
- See also: Arun B. Effects of myofascial release therapy on pain related disability, quality of sleep and depression in older adults with chronic low back pain. Int J Physiother Res 2014;2(1):318-23. — https://www.ijmhr.org/ijpr_articles_vol2_1/IJPR-2013-360.pdf
- See also: Duncan R. myofascial release hands-on guides for therapists. 1st ed. Florida, United States of America: Hum Kinet Inc 2014. — https://www.amazon.com/Myofascial-Release-Step-step-Hands/dp/1450444571
- See also: Thomas Scioscia M. Back Muscles and Low Back Pain. Spine-health. 2021. — https://www.spine-health.com/conditions/spine-anatomy/back-muscles-and-low-back-pain
- See also: Morán Esquerdo O, Arechabala I. Stretching Exercises Encyclopedia. Maidenhead: Meyer & Meyer Sport; 2013. — https://pdfroom.com/books/stretching-exercises-encyclopedia-by-oscar-moran-isabel-arechabala/andLVoyx2e3
- See also: Ohtsuki K et al. Comparison of the immediate changes in subjects with chronic lower back pain effected by lower back pain exercises and direct stretching of the tensor fasciae latae, the hamstring and the adductor magnus. J Phys Ther:2012;24(1):97-100.. — https://www.researchgate.net/publication/280080416
- See also: Raza S, Awan WA, Ghauri MW, Mahmood T, Abbas S. Effectiveness of spinal stabilization exercises with and without stretching of Latissimus dorsi Muscle in chronic mechanical low back pain. RMJ. 2020; 45(4): 857-862. — https://www.rmj.org.pk/?mno=130725
- See also: Sauer S, Biancalana M. Trigger point therapy for low back pain. New Harbinger Publications; 2010. — https://books.google.com.pk/books?hl=en&lr=&id=mSRpe9RS0uwC&oi=fnd&pg=PR5&dq=Trigger+Point+Therapy+for+Low+Back+Pain:+A+Self-treatment+Workbook+Sharon+Sauer,+Mary+Biancalana+-+Health+%26+Fitness+-+2010&ots=kgz3Z8_Jre&sig=vNYD1MIi_Pn2_Ke5iwdmaCkdzEI&redir_esc=y#v=onepage&q=Trigger%20Point%20Therapy%20for%20Low%20Back%20Pain%3A%20A%20Self-treatment%20Workbook%20Sharon%20Sauer%2C%20Mary%20Biancalana%20-%20Health%20%26%20Fitness%20-%202010&f=false